CLINICAL TRIAL: NCT04828720
Title: Clinical and Cytological Assessment of Platelet-Rich Fibrin and Topical Ozonated Oil in the Management of Palatal Wound Healing After Free Gingival Graft Harvest
Brief Title: Assessment of Platelet-Rich Fibrin and Topical Ozonated Oil in the Management of Palatal Wound Healing After Free Gingival Graft Harvest
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: October 6 University (Other)
Responsible Party: Principal Investigator, Asma Serag, lecturer of periodontology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000034
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Inadequately Attached Gingiva (Disorder)

STUDY DESIGN:
Intervention Model Description: In patients with inadequate zone of attached gingiva, treatment planned for FGGs to augment keratinized tissue dimensions in the mandibular incisor area.
Who Masked: Outcomes Assessor
Masking Description: opaque envelope
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRF group (Active Comparator): The PRF was prepared according to Choukroun et al. [5] immediately before surgery, a 10 ml blood sample was taken by venipuncture of the antecubital vein without anticoagulant. The tubes were centrifuged immediately by a dedicated centrifuge at 3,000 rpm for 10 minutes.
  A structured fibrin clot was produced by such preparation protocol in the middle of the tube, with the erythrocytes at the bottom and acellular plasma at the top. Following elimination of acellular plasma, a sterile scissors was used to separate the PRF from the erythrocytes. A membrane of PRF was formed by squeezing it gently between two pieces of gauze. Folding of the membrane was performed to achieve the required thickness (1.0 mm) with accurate trimming to match the palatal wound. The obtained membrane was then placed at the palatal donor site and compressed with gauze. Then, it was secured with 3-0 black plaited silk and a stent was placed.
  Interventions: Drug: ozonated oil
- Control group (Placebo Comparator): the palatal wounds in control group were managed by compressing the donor site with gauze and periodontal pack was placed. Patients in control group used a soft stent to protect the palatal donor wound site . Patients were instructed firmly not to shatter the stent for 1 week. The stent was removed and reseated only by the operator during the application of medications and collection of smears. One week postoperatively, the protective stents were discontinued.
  Interventions: Drug: ozonated oil
- ozonated group (Experimental): the palatal wound in ozanaited group will be painted by ozainated oil 2ml daily for 1 week, Patients used a soft stent to protect the palatal donor wound site . Patients were instructed firmly not to shatter the stent for 1 week. The stent was removed and reseated only by the operator during the application of medications and collection of smears. One week postoperatively, the protective stents were discontinued.
  Interventions: Drug: ozonated oil

INTERVENTIONS:
Drug: ozonated oil — All patients in ozone group were asked to visit the clinic on a daily basis through the first week and have their allocated therapeutic medication applied to their particular palatal donor site wounds. The wounds were coated with 2 ml ozonated oil per day, with a concentration of 15 µg of ozone/ml of olive oil. Moreover, palatal wounds in control group were managed by compressing the donor site with gauze and periodontal pack was placed. Patients in ozone group used a soft stent to protect the palatal donor wound site and to retain the tested oils in the post harvested palatal wounds. Patients were instructed firmly not to shatter the stent for 1 week. The stent was removed and reseated only by the operator during the application of medications and collection of smears. One week postoperatively, the protective stents were discontinued.

SUMMARY:
This randomized clinical trial was conducted to assess the effects of platelets-rich fibrin (PRF) and ozonated oil on the healing of palatal donor wound sites and the patient's morbidity after free gingival graft (FGG) harvesting

DETAILED DESCRIPTION:
Many surgical techniques have been suggested to enhance the width of keratinized tissue either by free gingival grafts (FGGs) or by sub-epithelial connective tissue grafts. FGG is easy to carry out and qualify the harvest of large quantities of connective tissues (CT). Contrariwise, it produces a site of secondary intention wound healing with discomfort and pain. Excessive post-operative morbidity has been reported in the literature as a possible complication of harvesting a FGG; different procedures with primary-intention healing have been proposed to overcome this problem.

The use of a platelet-rich fibrin (PRF) membrane to coat the fresh wound may accelerate the process of healing by providing a more stable rigid fibrin mesh, which is better than a blood clot and supplying a sustained release of growth factors promoting rapid hemostasis at the FGG donor site. PRF is a platelet concentrate obtained by inexpensive and simple procedure that does not need biochemical blood handling, it promotes efficient neovascularization, hastened wound closure and rapid cicatricial tissue remodeling through its three-dimensional fibrin meshwork. PRF owing its energizing effect on wound healing as it provides a superb scaffold for epithelialization and angiogenesis together with the presence of many growth factors such as platelet-derived growth factor (PDGF), epidermal growth factor and fibroblast growth factor (FGF).

Presently, most of researches in dental field using either ozone gas only, dissolved in water (ozonated water) or in plant oils such as olive oil (ozonated oil), focusing on its excellent antimicrobial efficacy, enhancement of wound healing in oral cavity without the possibility of drug resistance.

Oral wound healing is a dynamic process and complex phenomenon involving series overlapping stages of restoring tissue and cellular structures. Cellular and biochemical events in wound healing can be divided into several phases: inﬂammation, granulation tissue formation, matrix formation, re-epithelialization and tissue remodeling. Epithelial healing or re-epithelialization is an important process that involves the interactions between keratinocytes and extracellular matrix upon which cells migrate, proliferate and differentiate, hence restoring tissue function and structure. The rate of re-epithelization is considered as one of the criteria that reflect the influence of PRF and ozonated oil on healing of wound sites.

ELIGIBILITY:
Inclusion Criteria:

* (a) age ≥18 years and (b) healthy individuals without any systemic condition that might affect directly on the inflammatory status.

Exclusion Criteria:

* (1) patients with coagulation disorders, (2) severe psychiatric disorders, (3) heavy smokers, (4) patients wearing complete or partial denture that had any contact with the palate, (5) lactating or pregnant females and (6) no FGG harvested previously from the site.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
the Healing | assessed weekly for 1 month
  The healing assesed by healing index
  1- very poor. 5- excellent

SECONDARY OUTCOMES:
The Pain | after 24 hours and 1 week
  assessed by visual analogue scale (VAS)
cytological analysis | after 7, 14, 21 days and 2 months
  assess the re-epithelization and keratinization rate

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided